CLINICAL TRIAL: NCT01858285
Title: Genetics of Epilepsy and Related Disorders
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alissa D'Gama, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: X10-04-0197
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy; Epileptic Encephalopathy
Keywords: Epilepsy; Genetic
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA from whole blood, saliva, or buccal swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BCH Children's Rare Disease Cohort (CRDC): Individuals with epilepsy, onset at any age. Must be followed clinically at Boston Children's Hospital. Research trio-based exome and/or whole genome with CLIA confirmation of diagnostic findings. Exclusions include presence of existing genetic diagnosis or known cause for epilepsy, presence of structural brain malformation.
  Interventions: Genetic: Exome and/or whole genome sequencing

INTERVENTIONS:
Genetic: Exome and/or whole genome sequencing

SUMMARY:
Investigators at Boston Children's Hospital are conducting research in order to better understand the genetic factors which may contribute to epilepsy and related disorders. These findings may help explain the broad spectrum of clinical characteristics and outcomes seen in people with epilepsy.

DETAILED DESCRIPTION:
Many individuals with epilepsy experience seizures which respond well to treatment. Some types of epilepsy, however, are characterized by seizures which begin very early in childhood and are associated with severe intellectual and/or developmental disabilities. These conditions are often difficult to treat.

The investigators' research effort is focused on identifying genetic changes (known as "DNA variants") that cause epilepsy. By doing so the investigators hope to improve diagnosis and treatment for this epilepsy.

We have two specific aims:

1. Identifying genetic findings in patients with epilepsy and related disorders.
2. Correlating genetic findings with epilepsy phenotypes.

ELIGIBILITY:
inclusion: diagnosis of epilepsy, patient at Boston Children's Hospital exclusion: existing genetic diagnosis or known cause for epilepsy, structural malformation of the brain, not seen at Boston Children's Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with epilepsy. Age and epilepsy type variable.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-11; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identify new or existing pathogenic variants through exome and/or whole genome sequencing of individuals with epilepsy. | 10 years
  Use exome and/or whole genome sequencing to identify genetic variants. Detailed clinical information will be collected via medical records and patient questionnaire, as well as biological parents' exome sequencing to classify variants per ACMG guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Alissa D'Gama, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Epilepsy Genetics Program at Boston Children's Hospital website — https://www.childrenshospital.org/programs/epilepsy-genetics-program